CLINICAL TRIAL: NCT05674799
Title: NDPP-NextGen: A Clinical Trial to Reduce Intergenerational Obesity and Diabetes Risks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00108429; 1R01DK130900-01A1 (NIH)
Record Dates: First submitted 2022-11-21; First posted 2023-01-06 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-03

CONDITIONS: Overweight or Obesity
Keywords: Body mass index; Pre-conception; Diabetes Mellitus; Diet; Gestational diabetes; Neonatal adiposity; Maternal and Child Health; Overweight; Obese; Pregnancy; Randomized Control Trial; Weight; adverse maternal outcomes; Diabetes Prevention Program; glucose; gestational weight gain; lifestyle intervention; usual care; remote delivery; young women
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus; Diabetes, Gestational; Body Weight; Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to a 12-month lifestyle intervention promoting healthy diet and activity to reduce body weight (NDPP-NextGen), or usual care
Who Masked: Outcomes Assessor
Masking Description: Professional research assistants who will be collecting data and conducting the research visits will not be told if participants are in the treatment or control group, although this may be disclosed by the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Lifestyle (Experimental): Women in the Healthy Lifestyle group will be invited to attend the online NDPP-NextGen class which will cover how to eat healthy, be active, and lose weight before getting pregnant. The classes will be led by a trained Lifestyle Coach. Each class lasts about 1 hour. Classes initially meet about once a week (for the first 6 months), then twice a month (for the next 3 months), and then once a month (for the last 3 months). Classes will meet virtually through video-conference. Lifestyle coaches will also call participants in between classes to discuss how participants are doing, answer questions, and provide reminders for upcoming classes. Prior to the first class, women will also participate in a "pre-session" designed to increase NDPP engagement via discussion of diabetes risks and treatment options (i.e., clarify relevance) and motivational interviewing to resolve barriers.
  Interventions: Behavioral: NDPP-NextGen
- Healthy Women (No Intervention): Women in the Healthy Women group get a packet of information standardly given in OB clinics about how to be healthy before, during and after pregnancy.

INTERVENTIONS:
Behavioral: NDPP-NextGen — NDPP-NextGen will incorporate content on preconception/prenatal health into standard NDPP. Participants will be encouraged to make sustainable improvements in diet and activity, but without pre-set goals to better accommodate diverse, low-income populations. Upon pregnancy, recommendations will adjust to support appropriate GWG, breastfeeding, and postpartum weight loss. We will provide education on diet and activity during pregnancy/postpartum, including sufficient energy intake and exercise safety to support the growing fetus. NDPP-NextGen will include 3 strategies to better engage young women. (1) "Pre-sessions" to increase knowledge of diabetes risks, self-efficacy, and readiness to change using motivational interviewing techniques. (2) Delivering classes remotely (via phone- and video-conference) to facilitate participation regardless of inclement weather, dependent care, illness, transportation, etc. (3) Offering classes specially for young women to increase personal relevance.
  Arms: Healthy Lifestyle

SUMMARY:
The goal of this clinical trial is to test an enhanced version of the National Diabetes Prevention Program (NDPP-NextGen) that is tailored to young women in childbearing years. The investigators will recruit 360 women aged 18-39 years with overweight/obesity who are not currently pregnant, but likely to conceive within 24 months. Women will be randomized to NDPP-NextGen or a usual care control group. The NDPP-NextGen group will participate in the adapted NDPP online group class across 12 months, and the control group will get a packet of information about how to be healthy before, during and after pregnancy.

The main goals of the study are:

1. to assess effects of NDPP-NextGen on pre-pregnancy blood sugar and early pregnancy BMI
2. to assess effects of NDPP-NextGen on weight gain and behavioral outcomes during pregnancy
3. to explore effects of NDPP-NextGen on infant's percentage of fat tissue at birth

All participants will complete up to 4 research visits: baseline, conception, mid-pregnancy, and delivery. These visits will include:

1. Questionnaires about health, diet, activity, smoking, self-confidence, and depression
2. Body size measurements
3. Fasted blood draws

Participants will also be asked to weigh themselves weekly using home scales that are connected to the research database. At the delivery visit, investigators will measure the baby's body size and collect a cord blood sample.

DETAILED DESCRIPTION:
Intrauterine exposure to maternal overweight/obesity and diabetes transmits risks to offspring, triggering a disease cycle across generations. Over half of US women have overweight or obesity at conception and ~10% of pregnancies are affected by diabetes, exposing nearly 2 million infants each year. Prenatal lifestyle interventions are well-studied, yet begin too late to impact the critical period of conception and early pregnancy. Starting interventions before conception may be key to halting the disease cycle. However, prior research is limited, often lacks offspring outcomes (especially sensitive measures), includes mostly white and affluent participants, and has been challenged to identify women likely to conceive soon. Further research is needed on scalable strategies to improve maternal-child health during preconception and early pregnancy, especially for racial and ethnic minority or low-income women with disparately high prevalence of obesity and diabetes. The National Diabetes Prevention Program (NDPP) is a widely-disseminated lifestyle intervention to reduce weight and glycemia that has untapped potential to improve maternal-child health. From an implementation science perspective, the NDPP has greater potential impact than new interventions that are unlikely to be scaled up, even if efficacious. Denver Health has delivered the NDPP to >1600 adults since 2013, including >350 young women. Preliminary data shows that the NDPP may reduce peri-conceptional risks in diverse, low-income women. While limited engagement by younger women in the NDPP is a concern, strategies to increase engagement (motivational "pre-sessions", remote delivery, and classes specially for young women) are promising. For example, young women attended the 12-month NDPP for 64 days longer after receiving a pre-session, with 2.0 kg/m2 lower preconception BMI and 0.4% lower A1c in early pregnancy, than controls. To plan a preconception trial, the investigators developed a 2-step screening protocol to 1) use electronic health record data (e.g., contraceptive use) to identify women who are more likely to conceive by 24 months (36% vs. 13% for all young women), and 2) outreach to confirm current family planning to expect ≥60% conception, based on preliminary data showing that 73% conceived by 24 months if they endorsed intention to conceive or being sexual active without highly effective contraception. The investigators propose a randomized controlled trial of an enhanced NDPP (NDPP-NextGen) initiated before pregnancy to evaluate effects on maternal-child health. They will recruit 360 women aged 18-39 years with overweight/obesity who are likely to conceive within 24 months. Women will be randomized to NDPP- NextGen or a usual care control group. The specific aims are 1) to assess effects of NDPP-NextGen on peri- conceptional BMI and prenatal glycemia; 2) to assess effects of NDPP-NextGen on gestational weight gain and behavioral outcomes in pregnancy; and 3) to explore effects of NDPP-NextGen on neonatal adiposity and explanatory mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Established patient at Denver Health or Atrium Health Wake Forest Baptist
* Biologically female (inclusive of all gender identities)
* Aged 18-39 years
* English- or Spanish-speaking
* BMI ≥25 kg/m2 (≥23 kg/m2 if Asian race)
* Activities that lead to pregnancy in past 3 months
* Interested in pregnancy within 24 months, including:

  1. High interest (actively trying to conceive)
  2. General interest (not actively trying but wanting to become pregnant in the foreseeable future)
  3. Neutral interest (not planning pregnancy or using contraception for religious reasons)

Exclusion Criteria:

* Currently pregnant
* Non-gestational diabetes (type 1, type 2)
* Long-acting contraceptives (intrauterine device, implant, injection) with plans to continue for >1 year (barrier & short-acting hormonal contraception permitted given ease of discontinuing to facilitate pregnancy)
* Medical procedures (e.g., tubal ligation, hysterectomy) or conditions that impede pregnancy
* Documented infertility or unsuccessfully trying to conceive for ≥12 months
* Prior participation in the NDPP
* History of bariatric surgery
* Use of GLP-1s in last year
* Currently receiving clinical obesity treatment

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 403 (Estimated)
Dates: Start 2023-04-08 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
BMI in early pregnancy | 6-8 weeks gestation
  Height and weight will be measured and combined to report BMI at the post-conception research visit occurring at 6-8 weeks gestation.

SECONDARY OUTCOMES:
Glycemia in early pregnancy | 6-8 weeks gestation
  Fasting glucose

OTHER OUTCOMES:
Peri-conceptional BMI | Scale data will be pulled at 6-8 weeks gestation
  BMI at conception will be collected with cellular-enabled scales (BodyTrace®) that facilitate weekly at-home measurement to obtain weight closer to conception. Scales automatically transfer weights to a HIPAA-compliant database that is accessible only by the research team. Research staff will monitor for ≥1 transmitted weight each week, and provide prompts and assistance as needed. Investigators will average the two weights from before/after estimated date of conception to calculate approximate peri-conceptional BMI.
Rate and timing of gestational weight gain (GWG) | Scale data will be pulled weekly from time of conception up to delivery
  Primary method of collection will be through the use of home cellular scale weights. We will also abstract all weights from prenatal medical records as a secondary method to assess GWG. GWG will be analyzed as the difference from conception to delivery and gain within each trimester, adjusting for BMI at conception. We will also analyze GWG trajectories using linear mixed models with repeated measures drawn from the home scales and/or prenatal clinical weights. We will then classify women as having inadequate, appropriate, or excessive GWG based on BMI category, and analyze using logistic regression, again adjusting for BMI at conception.
A1C in early pregnancy | 6-8 weeks gestation
  Fasted blood draw
Glycemic status in early pregnancy | 6-8 weeks gestation
  Fasted blood draw to classify as normoglycemia, pre-diabetes, or type 2 diabetes at conception per American Diabetes Association definitions
Rate of gestational diabetes (GDM) in mid-pregnancy | 28-32 weeks gestation
  Abstracted from medical records
Diet quality | Baseline
  Diet will be assessed with 24-hour dietary recalls using the Automated Self-Administered system (ASA24). This system uses the USDA multiple-pass method to query all foods and supplements consumed in the prior 24 hours and produces daily and individual food estimates for macronutrients, micronutrients, and MyPyramid Equivalents (such as servings of vegetables, fruits, whole grains, solid fats, and added sugars).
Diet quality | 6-8 weeks gestation
  Diet will be assessed with 24-hour dietary recalls using the Automated Self-Administered system (ASA24). This system uses the USDA multiple-pass method to query all foods and supplements consumed in the prior 24 hours and produces daily and individual food estimates for macronutrients, micronutrients, and MyPyramid Equivalents (such as servings of vegetables, fruits, whole grains, solid fats, and added sugars).
Diet quality | 28-32 weeks gestation
  Diet will be assessed with 24-hour dietary recalls using the Automated Self-Administered system (ASA24). This system uses the USDA multiple-pass method to query all foods and supplements consumed in the prior 24 hours and produces daily and individual food estimates for macronutrients, micronutrients, and MyPyramid Equivalents (such as servings of vegetables, fruits, whole grains, solid fats, and added sugars).
Physical Activity | Baseline
  Assessed using the Pregnancy Physical Activity Questionnaire (PPAQ), while adjusting metabolic task equivalents for pregnancy. Investigators will calculate average activity intensity (sedentary to vigorous) and type (household, occupational, exercise, transportation) over the past 3 months at each collection point. Physical activity outcomes include daily minutes of sedentary, light, moderate, vigorous, household, occupational, exercise, transportation activity.
Physical Activity | 6-8 weeks gestation
  Assessed using the Pregnancy Physical Activity Questionnaire (PPAQ), while adjusting metabolic task equivalents for pregnancy. Investigators will calculate average activity intensity (sedentary to vigorous) and type (household, occupational, exercise, transportation) over the past 3 months at each collection point. Physical activity outcomes include daily minutes of sedentary, light, moderate, vigorous, household, occupational, exercise, transportation activity.
Physical Activity | 28-32 weeks gestation
  Assessed using the Pregnancy Physical Activity Questionnaire (PPAQ), while adjusting metabolic task equivalents for pregnancy. Investigators will calculate average activity intensity (sedentary to vigorous) and type (household, occupational, exercise, transportation) over the past 3 months at each collection point. Physical activity outcomes include daily minutes of sedentary, light, moderate, vigorous, household, occupational, exercise, transportation activity.
Smoking frequency | Baseline
  Participants will be asked about lifetime and recent (past 6 months) usage of cigarette and marijuana. Smoking outcomes include any smoking in pregnancy (binary) and number of cigarettes (total, trimester-specific).
Smoking frequency | 6-8 weeks gestation
  Participants will be asked about lifetime and recent (past 6 months) usage of cigarette and marijuana. Smoking outcomes include any smoking in pregnancy (binary) and number of cigarettes (total, trimester-specific).
Smoking frequency | 28-32 weeks gestation
  Participants will be asked about lifetime and recent (past 6 months) usage of cigarette and marijuana. Smoking outcomes include any smoking in pregnancy (binary) and number of cigarettes (total, trimester-specific).
Weight management self-efficacy | Baseline
  Assessed with the Weight Efficacy Lifestyle Questionnaire-Short Form (WEL-SF) on current confidence with weight management around negative emotions, availability, social pressure, physical discomfort, and positive activities. Weight management self-efficacy is a single score derived from the 8-item short form (range 0-72).
Weight management self-efficacy | 6-8 weeks gestation
  Assessed with the Weight Efficacy Lifestyle Questionnaire-Short Form (WEL-SF) on current confidence with weight management around negative emotions, availability, social pressure, physical discomfort, and positive activities. Weight management self-efficacy is a single score derived from the 8-item short form (range 0-72).
Weight management self-efficacy | 28-32 weeks gestation
  Assessed with the Weight Efficacy Lifestyle Questionnaire-Short Form (WEL-SF) on current confidence with weight management around negative emotions, availability, social pressure, physical discomfort, and positive activities. Weight management self-efficacy is a single score derived from the 8-item short form (range 0-72).
Rate of miscarriages | Through study completion, an average of 2 years
  Adverse maternal outcomes will be abstracted from medical records, and analyzed using logistic regression with consideration of a history of these conditions.
Rate of stillbirths | Through study completion, an average of 2 years
  Adverse maternal outcomes will be abstracted from medical records, and analyzed using logistic regression with consideration of a history of these conditions.
Rate of fetal deaths | Through study completion, an average of 2 years
  Adverse maternal outcomes will be abstracted from medical records, and analyzed using logistic regression with consideration of a history of these conditions.
Rate of pre-term births | Through study completion, an average of 2 years
  Adverse maternal outcomes will be abstracted from medical records, and analyzed using logistic regression with consideration of a history of these conditions.
Rate of pregnancy-induced hypertension | Through study completion, an average of 2 years
  Adverse maternal outcomes will be abstracted from medical records, and analyzed using logistic regression with consideration of a history of these conditions.
Rate of pre-eclampsia | Through study completion, an average of 2 years
  Adverse maternal outcomes will be abstracted from medical records, and analyzed using logistic regression with consideration of a history of these conditions.
Rate of eclampsia | Through study completion, an average of 2 years
  Adverse maternal outcomes will be abstracted from medical records, and analyzed using logistic regression with consideration of a history of these conditions.
Rate of cesarean delivery | Through study completion, an average of 2 years
  Adverse maternal outcomes will be abstracted from medical records, and analyzed using logistic regression with consideration of a history of these conditions.
Neonatal adiposity | At birth
  Percent of total mass that is fat mass, as measured by air displacement plethysmography using the PEA POD device
Maternal adiposity | Baseline
  Percent of total mass that is fat mass, as measured by air displacement plethysmography using the BOD POD device
Maternal adiposity | 6-8 weeks gestation
  Percent of total mass that is fat mass, as measured by air displacement plethysmography using the BOD POD device
Infant birthweight | At birth
  Medical records
Rate of macrosomia | At birth
  Infant birthweight >4000g. Abstracted from medical records
Rate of infants classified as large for gestational age (LGA) | At birth
  Infant birthweight >90th percentile. Abstracted from medical records
Rate of infants classified as small for gestational age | At birth
  Infant birthweight <10th percentile. Abstracted from medical records
Rate of infants with low birthweight | At birth
  Infant birthweight <2500g. Abstracted from medical records
Instances of fetal growth restriction | At birth
  Abstracted from medical records
Rate of infant birth trauma | At birth
  Abstracted from medical records
Rate of infant shoulder dystocia | At birth
  Abstracted from medical records
Rate of infant intensive care admission | At birth
  Abstracted from medical records
Rate of infants with a major congenital anomaly | At birth
  Abstracted from medical records
Rate of neonatal hypoglycemia requiring treatment | At birth
  Abstracted from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sauder, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No